CLINICAL TRIAL: NCT03386435
Title: The Effect of Remote Ischemic Preconditioning on the Postoperative Liver Function in Living Donor Hepatectomy: a Randomized Clinical Trial
Brief Title: The Effect of Remote Ischemic Preconditioning in Living Donor Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jun-Gol Song, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIPC_donor
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Tissue Donors; Liver Transplantation; Ischemia Reperfusion Injury
Keywords: remote ischemic preconditioning; liver donors
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: study group : remote ischemic preconditioning control group : none
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIPC (Experimental): intervention: RIPC groups receive remote ischaemic preconditioning after anaesthesia induction and before surgery started.
  Interventions: Procedure: remote ischemic preconditioning
- Control (No Intervention): In the control group, the same maneuver was applied but without cuff inflation.

INTERVENTIONS:
Procedure: remote ischemic preconditioning — Remote ischemic preconditioning was performed following anesthesia induction in donors. The protocol involves 3 cycles of 5-minute inflation of a blood pressure cuff to 200 mm Hg to one upper arm, followed by 5-minute reperfusion with the cuff deflated
  Other Names: RIPC
  Arms: RIPC

SUMMARY:
Liver transplantation is the gold standard treatment for patients with end-stage liver disease. Despite its outstanding success, liver transplantation still entails certain complications including ischemia-reperfusion injury. Remote ischemic preconditioning is a novel and simple therapeutic method to lessen the harmful effects of ischemia-reperfusion injury, however, the majority of remote ischemic preconditioning studies on hepatic ischemia-reperfusion injury have been animal studies. Therefore, our aim was to assess the effects of remote ischemic preconditioning on postoperative liver function in living donor hepatectomy.

DETAILED DESCRIPTION:
Liver transplantation(LT) is the gold standard treatment for patients with end-stage liver disease. In light of advancements in surgical techniques, immunosuppressive agents, and perioperative critical care, the overall 3-year survival of patients undergoing LT has exceeded 80%. Despite its outstanding success, LT still entails certain complications including ischemia-reperfusion injury (IRI).

IRI occurs when the blood supply to an organ or tissue is temporarily cut-off and then restored, and it is well-known as an underlying cause of primary non-function, biliary complications, and eventual graft loss after LT. Despite many attempts to ameliorate hepatic IRI, no definitive therapies have been established. In addition, the mechanisms of IRI remain largely unclear.

Remote ischemic preconditioning (RIPC) is a novel and simple therapeutic method to lessen the harmful effects of IRI. RIPC indicate that brief episodes of ischemia with intermittent reperfusion are introduced at a remote site, leading to systemic protection against subsequent insults as evinced on kidney, heart, liver, and other tissues. While RIPC has been shown to reduce hepatic IRI in several small animal studies, the beneficial effects of RIPC in hepatic IRI have been inconsistent. By far, the majority of RIPC studies on hepatic IRI have been animal studies; hence, there are limitations relating to the lack of human clinical trials.

Therefore, our aim was to assess the effects of RIPC on postoperative liver function in living donor hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Donors who plan to have living right hepatectomy for liver transplantation.
* age : between 18 to 60 years.

Exclusion Criteria:

* donors who plan to donate left lobe
* donors who plan to have laparoscopic right hepatectomy
* donors who cannot proceed remote ischemic preconditioning

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Gol Song, Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charlton MR. Improving long-term outcomes after liver transplantation. Clin Liver Dis. 2014 Aug;18(3):717-30. doi: 10.1016/j.cld.2014.05.011. PMID 25017085
- [Background] Foley DP, Fernandez LA, Leverson G, Chin LT, Krieger N, Cooper JT, Shames BD, Becker YT, Odorico JS, Knechtle SJ, Sollinger HW, Kalayoglu M, D'Alessandro AM. Donation after cardiac death: the University of Wisconsin experience with liver transplantation. Ann Surg. 2005 Nov;242(5):724-31. doi: 10.1097/01.sla.0000186178.07110.92. PMID 16244547
- [Background] Karp SJ, Johnson S, Evenson A, Curry MP, Manning D, Malik R, Lake-Bakaar G, Lai M, Hanto D. Minimising cold ischaemic time is essential in cardiac death donor-associated liver transplantation. HPB (Oxford). 2011 Jun;13(6):411-6. doi: 10.1111/j.1477-2574.2011.00307.x. Epub 2011 Apr 4. PMID 21609374
- [Background] Halladin NL. Oxidative and inflammatory biomarkers of ischemia and reperfusion injuries. Dan Med J. 2015 Apr;62(4):B5054. PMID 25872540
- [Background] Abu-Amara M, Yang SY, Quaglia A, Rowley P, Tapuria N, Seifalian AM, Fuller BJ, Davidson BR. Effect of remote ischemic preconditioning on liver ischemia/reperfusion injury using a new mouse model. Liver Transpl. 2011 Jan;17(1):70-82. doi: 10.1002/lt.22204. PMID 21254347
- [Background] Abu-Amara M, Yang SY, Quaglia A, Rowley P, de Mel A, Tapuria N, Seifalian A, Davidson B, Fuller B. Nitric oxide is an essential mediator of the protective effects of remote ischaemic preconditioning in a mouse model of liver ischaemia/reperfusion injury. Clin Sci (Lond). 2011 Sep;121(6):257-66. doi: 10.1042/CS20100598. PMID 21463257
- [Background] Gill R, Kuriakose R, Gertz ZM, Salloum FN, Xi L, Kukreja RC. Remote ischemic preconditioning for myocardial protection: update on mechanisms and clinical relevance. Mol Cell Biochem. 2015 Apr;402(1-2):41-9. doi: 10.1007/s11010-014-2312-z. Epub 2015 Jan 1. PMID 25552250
- [Background] Bjornsson B, Winbladh A, Bojmar L, Sundqvist T, Gullstrand P, Sandstrom P. Conventional, but not remote ischemic preconditioning, reduces iNOS transcription in liver ischemia/reperfusion. World J Gastroenterol. 2014 Jul 28;20(28):9506-12. doi: 10.3748/wjg.v20.i28.9506. PMID 25071345
- [Background] Hwang S, Lee SG, Lee YJ, Sung KB, Park KM, Kim KH, Ahn CS, Moon DB, Hwang GS, Kim KM, Ha TY, Kim DS, Jung JP, Song GW. Lessons learned from 1,000 living donor liver transplantations in a single center: how to make living donations safe. Liver Transpl. 2006 Jun;12(6):920-7. doi: 10.1002/lt.20734. PMID 16721780
- [Background] Jung KW, Kim WJ, Jeong HW, Kwon HM, Moon YJ, Jun IG, Song JG, Hwang GS. Impact of Inhalational Anesthetics on Liver Regeneration After Living Donor Hepatectomy: A Propensity Score-Matched Analysis. Anesth Analg. 2018 Mar;126(3):796-804. doi: 10.1213/ANE.0000000000002756. PMID 29256938
- [Background] Kim YK, Shin WJ, Song JG, Jun IG, Kim HY, Seong SH, Huh IY, Hwang GS. Effect of right ventricular dysfunction on dynamic preload indices to predict a decrease in cardiac output after inferior vena cava clamping during liver transplantation. Transplant Proc. 2010 Sep;42(7):2585-9. doi: 10.1016/j.transproceed.2010.04.041. PMID 20832549
- [Background] Rahbari NN, Garden OJ, Padbury R, Brooke-Smith M, Crawford M, Adam R, Koch M, Makuuchi M, Dematteo RP, Christophi C, Banting S, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Yokoyama Y, Fan ST, Nimura Y, Figueras J, Capussotti L, Buchler MW, Weitz J. Posthepatectomy liver failure: a definition and grading by the International Study Group of Liver Surgery (ISGLS). Surgery. 2011 May;149(5):713-24. doi: 10.1016/j.surg.2010.10.001. Epub 2011 Jan 14. PMID 21236455
- [Background] Selzner N, Rudiger H, Graf R, Clavien PA. Protective strategies against ischemic injury of the liver. Gastroenterology. 2003 Sep;125(3):917-36. doi: 10.1016/s0016-5085(03)01048-5. PMID 12949736
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Background] Hausenloy DJ, Erik Botker H, Condorelli G, Ferdinandy P, Garcia-Dorado D, Heusch G, Lecour S, van Laake LW, Madonna R, Ruiz-Meana M, Schulz R, Sluijter JP, Yellon DM, Ovize M. Translating cardioprotection for patient benefit: position paper from the Working Group of Cellular Biology of the Heart of the European Society of Cardiology. Cardiovasc Res. 2013 Apr 1;98(1):7-27. doi: 10.1093/cvr/cvt004. Epub 2013 Jan 19. PMID 23334258
- [Background] Robertson FP, Magill LJ, Wright GP, Fuller B, Davidson BR. A systematic review and meta-analysis of donor ischaemic preconditioning in liver transplantation. Transpl Int. 2016 Nov;29(11):1147-1154. doi: 10.1111/tri.12849. Epub 2016 Sep 20. PMID 27564598
- [Background] Imamura H, Kokudo N, Sugawara Y, Sano K, Kaneko J, Takayama T, Makuuchi M. Pringle's maneuver and selective inflow occlusion in living donor liver hepatectomy. Liver Transpl. 2004 Jun;10(6):771-8. doi: 10.1002/lt.20158. PMID 15162472
- [Background] Man K, Fan ST, Ng IO, Lo CM, Liu CL, Yu WC, Wong J. Tolerance of the liver to intermittent pringle maneuver in hepatectomy for liver tumors. Arch Surg. 1999 May;134(5):533-9. doi: 10.1001/archsurg.134.5.533. PMID 10323426
- [Background] Robertson FP, Fuller BJ, Davidson BR. An Evaluation of Ischaemic Preconditioning as a Method of Reducing Ischaemia Reperfusion Injury in Liver Surgery and Transplantation. J Clin Med. 2017 Jul 14;6(7):69. doi: 10.3390/jcm6070069. PMID 28708111
- [Background] Kanoria S, Jalan R, Seifalian AM, Williams R, Davidson BR. Protocols and mechanisms for remote ischemic preconditioning: a novel method for reducing ischemia reperfusion injury. Transplantation. 2007 Aug 27;84(4):445-58. doi: 10.1097/01.tp.0000228235.55419.e8. PMID 17713425
- [Background] Kanoria S, Robertson FP, Mehta NN, Fusai G, Sharma D, Davidson BR. Effect of Remote Ischaemic Preconditioning on Liver Injury in Patients Undergoing Major Hepatectomy for Colorectal Liver Metastasis: A Pilot Randomised Controlled Feasibility Trial. World J Surg. 2017 May;41(5):1322-1330. doi: 10.1007/s00268-016-3823-4. PMID 27933431
- [Background] Amador A, Grande L, Marti J, Deulofeu R, Miquel R, Sola A, Rodriguez-Laiz G, Ferrer J, Fondevila C, Charco R, Fuster J, Hotter G, Garcia-Valdecasas JC. Ischemic pre-conditioning in deceased donor liver transplantation: a prospective randomized clinical trial. Am J Transplant. 2007 Sep;7(9):2180-9. doi: 10.1111/j.1600-6143.2007.01914.x. PMID 17697262
- [Background] Franchello A, Gilbo N, David E, Ricchiuti A, Romagnoli R, Cerutti E, Salizzoni M. Ischemic preconditioning (IP) of the liver as a safe and protective technique against ischemia/reperfusion injury (IRI). Am J Transplant. 2009 Jul;9(7):1629-39. doi: 10.1111/j.1600-6143.2009.02680.x. Epub 2009 Jun 10. PMID 19519822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the donor group, adult (aged 18-60 years) liver donors scheduled for elective donor right hepatectomy from August 2016 to July 2017 at Asan Medical Center in Seoul, Korea, were screened for eligibility.
Groups:
- RIPC Group: received remote ischemic preconditioning
  remote ischemic preconditioning: transient brief episodes of ischemia at a remote site before a subsequent prolonged ischemia/reperfusion injury of the target organ
- Control Group: no intervention
Period: Overall Study
Arm/Group | RIPC Group | Control Group
Started | 80 | 80
Completed | 75 | 73
Not Completed | 5 | 7
Not completed — Protocol Violation | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIPC | Control | Total
Number analyzed (Participants) | 75 | 73 | 148
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 73 | 148
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 54 | 51 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 75 | 73 | 148
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 75 | 73 | 148
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (2.6) | 24.1 (2.7) | 23.9 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Postopera The Maximal Aspartate Aminotransferase Level Within 7 Postoperative Days
Description: The serial assessments of routine laboratory values were used as early markers for postoperative liver function. The maximal aspartate aminotransferase level within 7 postoperative days were assessed following RIPC in living donor hepatectomy.
Time Frame: within 7 days after operation
Measure: Mean (Inter-Quartile Range); unit: IU/L
Arm/Group | RIPC | Control
Number analyzed (Participants) | 75 | 73
IU/L | 145 [118.5 to 188] | 152 [129 to 180]

2. Primary Outcome: The Maximal Alanine Aminotransferase Level Within 7 Postoperative Days
Description: The serial assessments of routine laboratory values were used as early markers for postoperative liver function. The maximal alanine aminotransferase level within 7 postoperative days were assessed following RIPC in living donor hepatectomy
Time Frame: within 7 days after operation
Measure: Mean (Inter-Quartile Range); unit: IU/L
Arm/Group | RIPC | Control
Number analyzed (Participants) | 75 | 73
IU/L | 148 [120.5 to 197] | 152 [126 to 196]

3. Secondary Outcome: Number of Participants With Delayed Recovery of Liver Function
Description: The incidence of delayed recovery of hepatic function (DRHF) were used as surrogate parameters indicating the possible benefits of RIPC. DRHF was defined based on a proposal by the International Study Group of Liver Surgery, as follows: an impaired ability of the liver to maintain its synthetic, excretory, and detoxifying functions, which are characterized by an increased PT INR and concomitant hyperbilirubinemia (considering the normal limits of the local laboratory) on or after postoperative day 5. The normal upper limits of PT and bilirubin in our institutional laboratory were 1.30 INR and 1.2 mg/dL, respectively. If either the PT INR or serum bilirubin concentration was preoperatively elevated, DRHF was defined by an increasing PT INR and increasing serum bilirubin concentration on or after postoperative day 5 (compared with the values of the previous day).
Time Frame: postoperative 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | RIPC | Control
Number analyzed (Participants) | 75 | 73
Participants | 5 | 0

4. Secondary Outcome: Postoperative Liver Regeneration
Description: The postoperative liver regeneration index (LRI) at postoperative 1 month ) was used as surrogate parameters indicating the possible benefits of RIPC. The LRI was defined as [(VLR - VFLR)/VFLR)] × 100, where VLR is the volume of the liver remnant and VFLR is the volume of the future liver remnant. Liver volume was calculated by CT volumetry using 3-mm-thick dynamic CT images. The graft weight was subtracted from the total liver volume to define the future liver remnant.
Time Frame: 1 month
Measure: Mean (Inter-Quartile Range); unit: percentage of liver volume
Arm/Group | RIPC | Control
Number analyzed (Participants) | 75 | 73
percentage of liver volume | 83.3 [47.7 to 117.7] | 94.9 [61.4 to 131.2]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RIPC | Control
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/73
Other Adverse Events (participants affected / at risk) | 0/75 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT03386435/Prot_SAP_000.pdf